CLINICAL TRIAL: NCT04707690
Title: Intraurethral Laser Therapy for Stress Urinary Incontinence: A Randomized Sham - Controlled Clinical Study
Brief Title: IUL Study A Randomized Sham - Controlled Clinical Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: V1
Record Dates: First submitted 2021-01-12; First posted 2021-01-13 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Stress Urinary Incontinence
Keywords: Laser therapy; Stress urinary incontinence; intraurethral
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: Prospective randomized sham - controlled trial
Who Masked: Participant, Care Provider
Masking Description: Eligible patients will receive written and oral information about the study. After informed consent patients will be randomized into the intraurethral laser treatment group or sham laser group using the internet based program "randomizer", at a 1.1 ratio without stratification. Patients and the person performing the laser treatment will not aware of the treatment given. The laser devices can be used as a placebo laser blocking the laser beam with a plug.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intraurethral laser therapy (Active Comparator): Before treatment the vulva will be carefully inspected to rule out signs of infection or recent trauma. A local anesthetic fluid (Cathejell ®) will be applied to the urethral meatus. Before laser therapy, an intraurethral swab will be taken before treatment in order to determine the intraurethral microbiome.
  Vulvovaginal laser therapies will be performed with the non-ablative 2940 nm Er:YAG laser (Smooth XS, Fotona, Slovenia) in the Incontinence mode according to the manufacturer's guidelines and recommendations. The spot size (diameter of the laser beam) is 7 mm, with a pulse at a frequency of 1.6 Hz, and a fluence (laser energy delivered per unit area) of 5.0 to 10.0 J/cm2.
  Interventions: Device: Intraurethral laser therapy
- Intraurethral SHAM laser therapy (Placebo Comparator): Clinical examination and preparations will be identical to the intervention group. Sham laser treatments will be performed with the same laser and the same device. However, a specially designed placebo probe, which blocks the emission of radiation, will be used. Women will therefore receive no therapeutic laser treatment. Before treatment, a study assistant, who is aware of the study allocation, will prepare the laser with the placebo probe, which looks identically to the "normal" probe. The treating physician will not be aware of the study allocation and the type of probe in use.
  Interventions: Device: Intraurethral SHAM laser therapy

INTERVENTIONS:
Device: Intraurethral laser therapy — The laser will be applied according to the manufacturer's protocol. This includes a 2 step laser treatment using 2 different modes at 2 timepoints. The treatment takes about 15 minutes time.
  Other Names: Fotona smooth XS laser
  Arms: Intraurethral laser therapy
Device: Intraurethral SHAM laser therapy — The laser will be applied according to the manufacturer's protocol. This includes a 2 step laser treatment using 2 different modes at 2 timepoints. The treatment takes about 15 minutes time.
  Other Names: Fotona smooth XS laser
  Arms: Intraurethral SHAM laser therapy

SUMMARY:
Primary aim of the study is to compare the impact of SUI on the VAS (visual analogue scale) 3 months after laser therapy versus sham laser therapy.

DETAILED DESCRIPTION:
Background: Stress urinary incontinence (SUI) has a huge impact on the quality of life (QoL) in women and its treatment is challenging. Intraurethral laser may be an additional treatment option.

Study aim: The aim is to study the effectiveness of intraurethral laser therapy in women with SUI.

Design: randomized double blinded sham - controlled clinical study

Study population: women which have been diagnosed with SUI I-II°, aged between 18-80 years.

Study groups: Participants will be randomized (1:1), without stratification. The Intervention group will receive 2 treatments of intraurethral laser therapy and the Control group will receive 2 treatments of intraurethral SHAM laser therapy.

Sample size: A sample size of 20 women, 8 per group including a 20% Drop Out Rate, was calculated.

Primary outcome: impact of SUI on the VAS scale 3 months after laser therapy versus sham laser therapy.

Secondary study outcomes were defined as subjective SUI, objective SUI, QoL, treatment satisfaction, intraurethral microbiome, 3 months after laser therapy versus sham laser therapy.

ELIGIBILITY:
Inclusion Criteria:

* Female between 18 and 80 years
* Confirmed SUI through cough stress test within the last 24 months
* SUI I-II° for more than 6 months
* At least one incontinence episode per 24 hour period measured over three days according to a bladder diary
* Valsalva leak-point pressure (VLPP) ≤60 cm H2O
* Maximum cystometric capacity ≥250 mL
* No pelvic surgery within last 6 months (including prolapse repair, subjects who have residual or recurrent SUI following colposuspension or a sling procedure may be included in the study if the procedure was conducted at least 6 months prior to screening /baseline visit)
* BMI (body mass index) ≤35 kg/m2
* Willing to give informed consent and complete the follow up schedule

Exclusion Criteria:

* Active lower urinary tract infections (urethritis, cystitis or vaginitis)
* Three (3) or more cultured-proven bacterial urinary tract infection (UTI) in the last 12 months
* Detrusor overactivity on urodynamics
* Postvoiding residual (PVR) > 100 ml
* Previous urethral surgery (i.e. fistula or diverticula)
* Pelvic organ prolapse grade > 3 as defined by POP-Q and symptomatic
* Known polyuria (>3l/24h)
* Unevaluated macro hematuria
* Neurogenic bladder
* Evidence of dysplasia in a Pap smear (done in the last 24 months)
* Tumours of the Urinary tract
* Previous radiation or brachytherapy to treat pelvic cancer
* Uncontrolled diabetes
* Active herpes genitalis
* Pregnancy
* Vaginal delivery within 6 months prior to the Screening/Baseline Visit

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only females can participate in this study because it is led by gynecologists.
Enrollment: 20 (Estimated)
Dates: Start 2021-01-08 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Subjective symptoms of SUI | 3 months
  A visual analogue scale (VAS) is used for assessment for the subjective symptoms and improvement of SUI. Patients are asked to indicate the degree of their symptoms on a scle ranging from 0 (no symptoms) to 10 (worst possible symptoms).

SECONDARY OUTCOMES:
Degree of pain during laser therapy on a visual analogue scale (VAS) | 3 months
  Patients are asked to indicate the degree of pain during laser therapy on a visual analogue scale (VAS) ranging from 0 (no pain) to 10 (worst possible pain).
Subjective SUI | 3 months
  Subjective SUI as determined by the question "do you leak urine when coughing, sneezing or laughing" with the answer possibilities of "Yes" and "No".
Objective SUI | 3 months
  Objective SUI as determined by the cough stress test at 300ml bladder filling, which will either be positive or negative.
Patient Global Impression of Improvement | 3 months
  The PGI-I scales are robust and valid instruments to assess disease severity, bother and improvement after treatment in women and will be used to determine the Patient Global Impression of Improvement. The PGI-I consists of a 7-likert-scale with 7 being the worst bother.
Patient Global Impression of Severity | 3 months
  The Patient Global Impression of Severity (PGI-S) is a global index that may be used to rate the severity of a specific condition (in a single-state scale). The PGI-I scales are robust and valid instruments to assess disease severity, bother and improvement after treatment in women and will be used to determine the Patient Global Impression of Severity. The PGI scales are robust and valid instruments to assess disease severity, bother and improvement after treatment. The patient can choose from 4 answers including none, mild, moderate and severe.
Quality of Life using the Kings Health Questionnaire | 3 months
  The Kings Health Questionnaire was validated in women with stress urinary incontinence and assesses the impact of incontinence on quality of life. The eight subscales ("domains") scored between 0 (best) and 100 (worst). The Symptom Severity scale is scored from 0 (best) to 30 (worst); lower scores indicate better QoL. Success in terms of the study is defined as 10 points improvement on the total Kings Health Questionnaire score.
Pelvic floor symptoms | 3 months
  A validated self-administered pelvic floor questionnaire (Baessler) will be used to assess urogentinal symptoms. Questions regarding bladder (15), bowel (12), and sexual function (10), and pelvic organ prolapse symptoms (five) are grouped according to the physiological functions of the pelvic floor: bladder function, bowel function, prolapse symptoms, and sexual function domains. Quality of life measures and bothersomeness ratings were integrated into the four domains. Frequency, severity, and bothersomeness of pelvic floor symptoms are assessed using a four-point scoring system for most items in the questionnaire, apart from defecation frequency, bowel consistency, sufficient lubrication, and the reason for sexual abstinence. The lower the score the less pelvic floor symptoms the patients have.
Pad Weight | 3 months
  In regards to the one-hour stress pad weight test women are asked to drink 500 ml of sodium-free liquid in <15 min, then sit, walk for 30 min including climbing one flight of stairs. Afterwards the total amount of urine leaked is determined by weighing the pad. Lower weight means less urine loss.
Patient satisfaction with treatment/inpatient management | 3 months
  Patient satisfaction will be evaluated with the "Fragebogen zur Patientenzufriedenheit - ZUF-8". The German version of the original "Client Satisfaction Questionnaire-CSQ8", is a validated tool for measuring global patient satisfaction at the end of inpatient treatment. The ZUF-8 is an 8-items questionnaire to assess satisfaction in patients undergoing inpatient treatment. At 3 months treatment satisfaction will be assessed using an adopted version of the questionnaire. The lower the score, the higher is the patient satisfaction.
Microbiome | 3 months
  Extraction of archaeal/bacterial 16S rRNA gene using the Illumina MiSeq platform in order to determine the intraurethral microbiome

CONTACTS AND LOCATIONS:
Locations (1):
- Departement of Obstetrics and Gynecology, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No